CLINICAL TRIAL: NCT02124109
Title: The Genetic Basis of Acquired Heart Disease in Africa
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999914098; 14-HG-N098
Record Dates: First submitted 2014-04-25; First posted 2014-04-28 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Rheumatic Heart Disease; Rheumatic Fever; Endomyocardial Fibrosis; Acquired Heart Disease
Keywords: Rheumatic Heart Disease
MeSH Terms: conditions — Rheumatic Heart Disease; Rheumatic Fever; Endomyocardial Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Control: Control group
- rheumatic heart disease: Patients with rheumatic heart disease

SUMMARY:
Background:

- An acquired heart disease is one that a person gets after they are born. Two of these are rheumatic heart disease (RHD) and endomyocardial fibrosis (EMF). They are found more commonly in people who live in Africa than in other places in the world. Researchers want to learn more about these diseases. They especially want to know what role genes and other factors play in them.

Objective:

- To identify genetic risk factors for RHD and EMF in sub-Saharan Africa.

Eligibility:

* Children and adults with RHD or EMF.
* Healthy volunteers over age 10.

Design:

* Participants will come from existing study groups in Uganda and Nigeria.
* Participants may be required to provide a sample of their DNA. They will do this with either a blood or saliva sample or a swab of the mouth.
* Collected samples will be labeled with a code and sent to a lab in the United States for analysis. Remaining portions of participants samples will be stored for an unlimited period of time. They may be used in future studies.
* Some genetic and health information from participants might be placed into one or more scientific databases.
* Participant names and identifying information will be kept private. But there is a small chance someone could trace them from their genetic information.

DETAILED DESCRIPTION:
Recent advances in genomic techniques are making possible a new wave of genetic discovery in many complex diseases. However, the genetic risk factors for two forms of acquired heart disease that are particularly common in Africa - rheumatic heart disease (RHD) and endomyocardial fibrosis (EMF) remains unknown. In this application, we propose to evaluate genetic risk factors for rheumatic heart disease (RHD) and endomyocardial fibrosis (EMF). A number of factors should facilitate the identification of genetic risk variants underlying the two conditions. First, both forms of acquired heart disease are endemic to sub-Saharan Africa (SSA). Second, affected patients and those who do not develop the conditions share a common environment. Finally, the availability of high density SNP arrays to capture common and rare variation makes the characterization of genomic variation better than ever. Patients will be enrolled at the Uganda Heart Institute in Kampala, Uganda, and at the College of Medicine, University of Lagos, Nigeria, with the potential to include other African sites. Genomic studies will be done at the NIH.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Rheumatic Heart Disease:

Patients with a definite diagnosis of rheumatic heart disease based on the 2006 World Health Organization/National Institutes of Health Joint Criteria (http://www.niaid.nih.gov/topics/strepThroat/Documents/groupasequelae.pdf) controls who do not meet this criteria. The diagnosis will be made by a cardiologist on our team. The method of screening and recruitment will be specific to each of our two sites: Uganda Heart Institute and University of Lagos, Nigeria.

-Uganda Heart Institute:

--recruitment will be conducted from an existing cohort of patients initially recruited by members of our team from 21 randomly selected

schools in Uganda. Participants meeting the criteria noted above for RHD will be considered cases and those who do not will be considered controls. Additionally, parents will be invited to participate as controls. For controls, only children over age 10 will be considered as this increases the likelihood of exposure

to S. pyogenes. The initial study was approved by the institutional review boards of the Children s National Medical Center (Washington,D.C.), Makerere University (Kampala, Uganda), and the

Ugandan Ministries of Health and Education

* University of Lagos:

  --This program will be modeled after the Uganda program. Participants will be screened for RHD at the College of Medicine or at randomly selected schools. Participants meeting criteria for RHD will be consented as cases and those negative for RHD will be consented as controls. Additionally, parents will be invited to participate as controls. For controls, only children over age 10 will be considered as this increases the likelihood of exposure to S. pyogenes
* Endomyocardial Fibrosis (EMF):

  * Cases: the study will include patients with a diagnosis of EMF based on echocardiography, history, and physical exam performed by cardiologist;on our team Over 50 patients have been identified at the Uganda Heart Institute with EMF and will be contacted for study participation; additionally, newly diagnosed patients at the Uganda Heart Institute will be offered participation.
  * Controls: Geographic and age matched controls will be used for association study. Controls will be disease free, based on above criteria. We will exclude controls less than 15 years of age based on disease peak around age 10. Controls will be selected from those being screening for RHD

EXCLUSION CRITERIA:

-Anyone unwilling to provide informed consent (for themselves as adults, or on behalf of their children as minors) or assent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with rheumatic heart disease@@@
Sampling Method: Non-Probability Sample
Enrollment: 736 (Actual)
Dates: Start 2014-04-03 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2020-02-06 (Actual)

PRIMARY OUTCOMES:
Extension of study | ongoing
  Extend our previous epidemiological studies of RHD in Ugandan schoolchildren (Beaton et al 2012) by conducting a similar study ofRHD in Nigerian children

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Kruszka, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (2):
- University of Lagos, Lagos, Nigeria
- Mulago Hospital, Kampala, Uganda